CLINICAL TRIAL: NCT06050512
Title: Phase I/II Trial of Mezigdomide Plus Ixazomib and Dexamethasone for Relapsed and Refractory Multiple Myeloma
Brief Title: Mezigdomide Plus Ixazomib and Dexamethasone for Relapsed and Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closure of trial per BMS
Sponsor: Kathleen Dorritie (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Kathleen Dorritie, Assistant Professor Hematology/Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-200
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Relapsed and Refractory Multiple Myeloma
Keywords: Bi-specific T-cell engaging antibodies (BITE); cereblon E3 ligase modulator (CELMoD); cereblon-mediated ubiquitination; cellular transcription factors (Ikaros and Aiolos)
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — ixazomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase l: Mezigdomide + Ixazomib + Dexamethasone (Experimental): Dose level -2: Mezigdomide: 0.3 mg daily on days 1-21 of a 28-day schedule; Ixazomib: 2.3 mg PO weekly on days 1, 8 and 15 of a 28-day schedule; Dexamethasone: 40 or 20 mg on days 1, 8, 15 and 22 Dose level -1: Mezigdomide: 0.6 mg daily on days 1-21 of a 28-day schedule; Ixazomib: 2.3 mg PO weekly on days 1, 8 and 15 of a 28-day schedule; Dexamethasone: 40 or 20 mg on days 1, 8, 15 and 22 Dose level 0 (Starting dose): Mezigdomide: 0.6 mg daily on days 1-21 of a 28-day schedule; Ixazomib: 3.0 mg PO weekly on days 1, 8 and 15 of a 28-day schedule; Dexamethasone: 40 or 20 mg on days 1, 8, 15 and 22 Dose level +1: Mezigdomide: 1.0 mg daily on days 1-21 of a 28-day schedule; Ixazomib: 3.0 mg PO weekly on days 1, 8 and 15 of a 28-day schedule; Dexamethasone: 40 or 20 mg on days 1, 8, 15 and 22 Dose level +2: Mezigdomide: 1.0 mg daily on days 1-21 of a 28-day schedule; Ixazomib: 4.0 mg PO weekly on days 1, 8 and 15 of a 28-day schedule; Dexamethasone: 40 or 20 mg on days 1, 8, 15 and 22
  Interventions: Drug: Mezigdomide; Drug: Ixazomib; Drug: Dexamethasone
- Phase ll (RP2D): Mezigdomide + Ixazomib + Dexamethasone (Experimental): Mezigdomide: RP2D daily on days 1-21 of a 28-day schedule Ixazomib: RP2D PO weekly on days 1, 8 and 15 of a 28-day schedule Dexamethasone: RP2D on days 1, 8, 15 and 22
  Interventions: Drug: Mezigdomide; Drug: Ixazomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Mezigdomide — Mezigdomide (MEZI), a novel oral CELMoD® agent with enhanced tumoricidal and immune-stimulatory effects compared to immunomodulatory drugs (IMiDs®), induces maximal degradation of Ikaros and Aiolos, leading to increased apoptosis in myeloma cells.
  Other Names: CC-92480; MEZI
Drug: Ixazomib — Ixazomib, a second-generation proteasome inhibitor, is used primarily in the treatment of multiple myeloma. This activity outlines the mechanism of action, indications, and contraindications for ixazomib as a valuable agent for treating multiple myeloma.
  Other Names: NINLARO®
Drug: Dexamethasone — Corticosteroids, such as dexamethasone and prednisone, are an important part of the treatment of multiple myeloma. They can be used alone or combined with other drugs as a part of treatment. Corticosteroids are also used to help decrease the nausea and vomiting that chemo might cause.
  Other Names: Dex

SUMMARY:
Multiple myeloma (MM) is the second most common hematologic malignancy with an estimated annual incidence of nearly 35,000 cases. While still considered an incurable disease, new treatments have improved outcomes dramatically over the last two decades. Around the turn of the millennium, classical cytotoxic chemotherapy and radiation were the only available treatment modalities and median OS was estimated at 2-3 years. Currently, there are now 17 FDA-approved anti-myeloma agents and median OS is approaching 10 years. More recently, next generation cellular and immune therapies are demonstrating unprecedented efficacy in highly refractory patients with otherwise a very short life expectancy. In this study, the starting dose of ixazomib will be reduced to 3mg, as this is the first FDA-recommended dose recommendation (from 4mg). The starting dose of mezigdomide will be 0.6mg. Frequent toxicity and AE monitoring as outlined in this trial (weekly in C1, every 2 weeks in C2-C4) asserts maximization of patient safety. Dexamethasone (DEX) will be dosed at 40mg weekly in patients < 75 years old and 20mg for patients > 76 years old. Additionally, the staring dose of DEX may be reduced to 20mg in any patient, per study provider discretion, based on several factors such frailty, prior adverse side effects or existing comorbidities.

DETAILED DESCRIPTION:
Mezigdomide is a novel cereblon E3 ligase modulator (CELMoD). It is an oral small-molecule compound that potentiates the cereblon-mediated ubiquitination of key cellular transcription factors (Ikaros and Aiolos), which ultimately results in multiple myeloma cell death and other immunomodulatory activity. Mezigdomide has demonstrated acceptable safety in two phase I clinical trials in combination with DEX as a "doublet," and as a "triplet" in combination with bortezomib and DEX. Early estimates of efficacy are high compared to historical date: 55% ORR in combination with DEX in a highly pre-treated and refractory patient population, and 75% in combination with bortezomib. By comparison, the most recent oral therapy approved by the FDA for RRMM was Selinexor, which demonstrated a 25% ORR in patients who received a median of 7 prior lines of therapy and 100% of whom were refractory to a PI, IMID and DARA. This comparison serves as very exploratory estimate as no conclusions can be drawn from cross-trial comparisons, especially with very small patient populations. While important efficacy measures such overall survival, progression-free survival and duration of response are maturing, these estimates suggest mezigdomide could be an efficacious, oral treatment option for patients with RRMM.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status < 2
* Patients must have a confirmed diagnosis of multiple myeloma and have received 1-3 prior lines of therapy and must be:
* Exposed to a proteasome inhibitor, IMiD, and anti-CD38 antibody prior to enrollment. Patients must have measurable evidence of multiple myeloma defined as one of the following:

  * Serum M protein ≥ 0.5 g/dL
  * Abnormal free light chain ratio, provided involved light chain is >10mg/dL
  * Urine M protein ≥ 200 mg/24 hours
* Hematologic laboratory parameters of:

  * Absolute neutrophil count (ANC) > 1,000/mm3
  * Hemoglobin > 8g/dL
  * Platelet count > 75,000/μL if plasma cells account for < 50% bone marrow
  * Nucleated cells and > 50,000/μL if plasma cells account for > 50% of bone marrow nucleated cells
* Non-hematologic laboratory parameters of:

  * Total Bilirubin of < 2 times the upper limit of normal
  * ALT and AST < 3 times the upper limit of normal
  * Corrected serum calcium >13 mg/dL
* Estimated creatinine clearance (CrCl) of ≥ 45 mL/min, calculated using the formula of Cockroft and Gault (may need adjusted per mezigdomide pharmacokinetic report)
* Access to ixazomib
* Females of childbearing potential (FCBP) must:

  o Have two negative pregnancy tests prior to starting study treatment and agree to ongoing pregnancy testing during the course of the study, and after end of study treatment.
* All male and female participants must follow all requirements defined in the pregnancy prevention plan

Exclusion Criteria:

* Central Nervous system involvement of multiple myeloma
* Plasma cell leukemia defined as clonal plasma cells constituting > 20% of peripheral leukocyte differential
* Waldenstrom's Macroglobulinemia, POEMS syndrome or Light Chain (AL) AmyloidosisF
* Prior refractoriness to a proteasome inhibitor (bortezomib, carfilzomib, ixazomib), defined as documented progression within 60 days of a PI-containing regimen
* Prior intolerance of ixazomib
* Prior exposure to mezigdomide
* Females with positive pregnancy test during screening or females who wish to become pregnant
* Unwillingness to strictly adhere to the Pregnancy Prevention Plan
* Concomitant or recent (within 2 weeks of starting study therapy) use of strong CYP3A modulators and proton pump inhibitors (PPIs)
* Active cardiopulmonary conditions including documented myocardial ischemia within 6 months, unstable angina, congestive heart failure (New York Heart Association class III or IV), uncontrolled arrythmias, Grade 3 conduction block without a pacemaker, uncontrolled hypertension, baseline QTc >470ms or chronic obstructive pulmonary disease with FEV1 <50%
* Any other malignancy diagnosed within 2 years of enrollment with documented or presumed residual disease, excluding non-melanomatous skin cancer if completely resected
* Active bacterial or fungal infection requiring antimicrobial therapy (not standard prophylactic prophylaxis)
* HIV, chronic or active hepatitis B, or active hepatitis A or C
* Unwillingness to adhere to antithrombotic and antiviral prophylaxis
* Major surgery within 30 days of enrollment
* Radiotherapy within 14 days of initiating study treatment
* Known allergy to any study compounds (mezigdomide, ixazomib)
* Intolerance of dexamethasone
* Documented gastrointestinal disease resulting reduced absorption of oral medications
* Grade > 3 neuropathy
* Active participation in another clinical trial or recent participation within 1 month of enrollment
* Any medical or psychiatric condition interfere with the patient's ability to tolerate or complete this treatment protocol, as determined by principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Phase l: Recommended Phase II Dose (RP2D) | Up to 17 months
  Dose-limiting toxicity (DLT) per adverse events as defined using National Cancer Institute (NCI) CTCAE v5.0. Hematologic DLTs: Grade 4 neutropenia < 500/μL for more than 5 days, Grade 3 neutropenia with fever > 38.3°C (one time) or fever > 38.0°C sustained for one hour, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with bleeding; Non-Hematologic DLTs: Grade 3 diarrhea lasting >3 days (not recovering to < grade 2) despite supportive care, Grade 3 nausea or vomiting >3 days (not recovering to < grade 2) days despite supportive care, Grade 3 fatigue lasting >7 days (not recovering to < grade 2) days despite supportive care, Grade 4 diarrhea, Grade 4 nausea or vomiting, Allergic reaction or hypersensitivity if unable to be corrected to <grade 1 within 48 hours, Any other non-hematologic grade >3 toxicity for which there is not a clear alternative explanation; General: dose modification or delay of mezigdomide or ixazomib during cycle 1 due to treatment related toxicity.
Phase ll: Overall Response Rate (ORR) | Up to 36 months
  Preliminary efficacy of mezigdomide when given in combination with ixazomib and dexamethasone as estimated by ORR, as defined by the International Myeloma Working Group (IMWG) response criteria. This will be expressed as the proportion of patients who achieve complete response (CR) or partial response (PR). CR is defined as negative serum and urine M-protein immunofixation (IF), along with the presence of < 5% plasma cells (PCs) in bone marrow (BM) biopsy. PR is defined as ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours.

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events | Up to 36 months
  Incidence and severity of adverse events AEs, as defined by the NCI-Common Terminology Criteria for Adverse Events v5.0, tabulated by type, grade and relatedness to treatment for each dose level achieved in the study and overall.
Depth of Response | Up to 36 months
  Depth of Response will be measured as the proportion of participants in each category, given IMWG Uniform Response Criteria at each dose level and overall.
Duration of Response (DOR) | Up to 36 months
  The time from the date of the earliest documented response (PR, VGPR, CR or sCR) to the earliest date of disease progression or death, whichever occurred first. Disease progression will be determined by the investigator per IMWG Uniform Response Criteria.
Progression-free Survival (PFS) | Up to 36 months
  The time from the date of first treatment to the earliest date of disease progression or death, whichever occurred first. Disease progression will be determined by the investigator per IMWG Uniform Response Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Dorritie, MD, Principal Investigator — UPMC Hillman Cancer Center

IPD SHARING:
Plan to Share IPD: No